CLINICAL TRIAL: NCT05595395
Title: The Enteral Resuscitation In Intensive Care (ERI) Pilot- Study: Enteral Versus Intravenous Fluid Administration in the Treatment of Critically Ill Patients: a Randomized Controlled Pilot Trial
Brief Title: The Enteral Resuscitation In Intensive Care Pilot- Study
Acronym: ERI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Collaborators: Klinik Favoriten (Other)
Responsible Party: Principal Investigator, Assoc. Prof. Dr. Manfred Hecking, MD PhD, Principal Investigator, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EK Nr. 1790/2020
Record Dates: First submitted 2022-10-22; First posted 2022-10-27 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Electrolyte Imbalance; Volume Overload; Hyperosmolality
Keywords: Fluid Therapy; Critical Care; Prospective Studies; Pilot Project
MeSH Terms: conditions — Edema | interventions — Infusions, Intravenous

STUDY DESIGN:
Intervention Model Description: Prospective, explorative, multicenter, randomized, parallel group, open-label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intravenous Fluid Arm (Placebo Comparator): In Group 1 (Standard of practice/intravenous fluid group) no enteral administration of fluid other than enteral nutrition is going to be allowed. Intravenous fluid administration is going to be administered at the discretion of the physician in charge and "Elomel isoton" is going to be the fluid of choice.
  Interventions: Drug: Intravenous Infusion
- Enteral Fluid Arm (Active Comparator): In Group 2 (Test practice/enteral fluid group) enteral fluid administration is going to be the primary mode of administration. Intravenous fluid administration can be performed by physicians at their own discretion. Primary enteral fluid administered is going to be tap water, intravenous fluid of choice is going to be "Elomel isoton".
  Interventions: Drug: Enteral Dose Form

INTERVENTIONS:
Drug: Enteral Dose Form — In this intervention arm, fluid substitution is primarily done via enteral administration. The used substance for enteral fluid administered is going to be tap water. Intravenous fluid of choice is going to be "Elomel isoton".
  Arms: Enteral Fluid Arm
Drug: Intravenous Infusion — In this intervention arm, fluid substitution is primarily done via intravenous administration. The used substance for intravenous fluid administered is going to be "Elomel isoton".
  Arms: Intravenous Fluid Arm

SUMMARY:
The purpose of this pilot study is to overcome the limited evidence on enteral fluid administration in intensive care medicine and to generate data for further hypothesis generation in an exploratory setting. This trial is a prospective, multicenter, randomized, parallel group, open-label study to compare the current standard of practice, the intravenous fluid administration, with a more physiological approach, the enteral fluid administration, in critically ill patients.

DETAILED DESCRIPTION:
Introduction: The effectiveness and safety of enteral fluid administration in critically ill patients remains unclear. Existing evidence regarding this topic is scarce, but suggests that enteral fluid administration is a safe route of administration. To our knowledge no randomized controlled trial has been conducted investigating this topic.

Objectives: The aim of this pilot study is to gather evidence on the impact of enteral fluid replacement on clinical, laboratory and outcome parameters in intensive care patients in order to plan a subsequent larger randomized controlled trial. Clinical outcomes indices evaluated are regurgitation, thirst, serum sodium, mortality, length of mechanical ventilation arterial pressure, urinary volume, body weight, edema, intra-abdominal pressure), changes in bioimpedance spectroscopy-derived markers, fluid overload, renal function tests, liver function tests and SOFA-Scores.

Methods: The trial is a prospective, multicenter, randomized, parallel group, open-label study. Patients are going to be recruited and randomized at 3 separate internal medicine intensive care units in Vienna, Austria. A total of 64 patients will be recruited and randomized to receive enteral fluid administration via nasogastric tube or intravenous administration only. Daily visits and evaluation of clinical and radiological fluid status is performed by the attending physician. Regular study visits with Bioimpedance spectroscopy measurements (BIS) to evaluate fluid status are going to be performed

Results and conclusions: The ERI study will provide data on potential outcome parameters to plan a subsequent larger randomized control trial for patients receiving enteral fluid therapy in intensive care medicine.

Ethics and dissemination: The trial is performed in accordance with the Declaration of Helsinki. It subscribes to the principles outlined in the most recent version of the International Conference on Harmonization on Good Clinical Practice. Approval was obtained from the ethics committee of the Medical University of Vienna (EK number 1790/2020). The study has also been registered in a public clinical trial database (EudraCT Identifier Number 2018-002447-29, clinicaltrialsregister.eu).

ELIGIBILITY:
* Inclusion criteria:

  * Patient intubated within the last 72h
  * Age >18 years
  * Expected required fluid volume may not exceed 4 mL/kg/h (permanently, during at least 24 hours).
  * Negative pregnancy test in female patients of childbearing potential
  * Informed consent. For patients that are temporarily unable to consent a
  * subsequent informed consent must be provided.
* Exclusion criteria:

  * Evidence of severe gastrointestinal disease defined as

    * Gastrointestinal Failure with > 3 symptoms (see below) or
    * Lactate >3mmol/L when mesenterial ischemia is a probable cause
    * Clinical signs of intra-abdominal hypertension and an increase of intra-abdominal pressure of >20 mmHg.
  * Patients who cannot receive early enteral nutrition due to conditions such as prone positioning in consequence of conditions such as acute respiratory distress syndrome
  * Pregnancy
  * Abdominal surgery in the last 3 months (unless all involved physicians, study investigators and caretaking doctors agree that the surgical event does not constitute a limitation for enteral fluid administration)
  * Postoperative patients with consecutive admission to ICU
  * Extracorporeal Kidney-Replacement Therapy before intubation
  * At the discretion of the Investigator

Symptoms of Gastrointestinal Failure:

* Absent bowel sounds
* Bowel distension
* Vomiting/regurgitation volume >500 ml
* GI bleeding
* Diarrhoea (liquid stool >3 times a day)
* Distended stomach on ultrasound examination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2023-02-13 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Regurgitation | From the moment of intubation to extubation.
  Incidence and extent of regurgitation via the stomach/jejunal probe
Sodium/Osmolality | From the moment of intubation to extubation.
  Differences of serum sodium and serum osmolality
Thirst | On the last study visit (day of extubation)
  Thirst on a zero to 10 numeric rating scale (NRS; worst = 10)
Days on ventilation | From the moment of intubation to extubation.
  Days on ventilation
30-day mortality | From the moment of intubation until 30 days after intubation
  30-day mortality

SECONDARY OUTCOMES:
Kidney Failure | From the moment of intubation to extubation.
  Incidence and extent of kidney failure as well as kidney function
SOFA-Score | From the moment of intubation to extubation
  Differences of Sequential Organ Failure Assessment (SOFA) Scores of patients. This score includes PaO2 [mmHg], FiO2 [%], mechanical ventilation [Yes/No], Platelets [/µL], Glascow Coma Scale, Bilirubin [mg/dL], Mean arterial pressure OR administration of vasoactive agents required and creatinine [mg/dL]. The score ranges from 0=best to 24=worst.
BCM | From the moment of intubation to extubation
  Differences in fluid volume status including Bioimpedance spectroscopy measurements (BIS) using Body Composition Monitor (BCM)

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Hecking, M.D., Principal Investigator — Medical University of Vienna, Department of Nephrology and Dialysis
Locations (2):
- Austria (2):
  - Klinik Favoriten, Vienna
  - Department of Internal Medicine III, Division of Nephrology and Dialysis, Medical University of Vienna, Austria, Vienna

IPD SHARING:
Plan to Share IPD: No